CLINICAL TRIAL: NCT00003583
Title: A Phase II Trial Using Amifostine as a Chemo/Radio Protective Agent in the Treatment of Limited Stage Small-Cell Lung Cancer
Brief Title: Amifostine to Prevent Side Effects in Patients Who Are Receiving Chemotherapy and Radiation Therapy for Limited-Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Florida (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000066651; UF-G-97120405; ALZA-97-033-ii; NCI-V98-1475
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2006-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Radiation Toxicity
Keywords: limited stage small cell lung cancer; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Radiation Injuries | interventions — Amifostine; Cisplatin; Etoposide; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Drugs such as amifostine may protect normal cells from the side effects of chemotherapy and radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of amifostine to prevent side effects in patients who are receiving chemotherapy and radiation therapy for limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the reduction in toxicities by combining amifostine with cisplatin, etoposide, and radiotherapy in patients with limited stage small cell lung cancer. II. Evaluate the response rate to this combination by these patients. III. Evaluate the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive cisplatin IV on day 1 and etoposide IV daily on days 1-3. This course is repeated every 3 weeks for a total for 4 courses. Patients also receive concurrent radiotherapy 5 days per week for 5.5 weeks starting with the first course of chemotherapy. Patients receive amifostine IV over 15 minutes 15-30 minutes prior to each dose of chemotherapy on days 1-3. Patients are followed at 6 and 12 weeks, then every 3 months for 9 months, every 6 months for 1 year, and then until death.

PROJECTED ACCRUAL: There will be 20 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed limited stage small cell lung cancer Primary tumor must be evaluable radiographically

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 Life expectancy: At least 3 months Hematopoietic: WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT and SGPT less than 2 times normal Renal: Creatinine less than 1.5 mg/dL Other: No concurrent active infection No prior malignancy except squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: Dean L. McCarley, MD, Study Chair — Veterans Affairs Medical Center - Gainesville
Locations (1):
- University of Florida - Gainesville, Gainesville, Florida, United States